CLINICAL TRIAL: NCT04256798
Title: PErioperative Respiratory Care and Outcomes for patieNts Undergoing hIgh Risk abdomiNal Surgery: A 2x2 Factorial, International Pragmatic Randomised Controlled Trial Across Low and Middle-income Countries
Brief Title: Perioperative Respiratory Care and Outcomes for Patients Undergoing High Risk Abdominal Surgery
Acronym: PENGUIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RG_19-223
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Infection; Pneumonia; Surgical Site Infection; Wound Infection; Surgical Wound Infection; Postoperative Complications; Anesthesia; Communicable Disease; Pathologic Processes; Perioperative Complication; Chlorhexidine; Laparotomy
MeSH Terms: conditions — Infections; Pneumonia; Surgical Wound Infection; Wound Infection; Postoperative Complications; Communicable Diseases; Pathologic Processes | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mouthwash and liberal oxygen during surgery (Experimental): Pre-surgical mouthwash with 0.2% chlorhexidine gluconate in combination with 80-100% FiO2 during surgery.
  Interventions: Drug: Chlorhexidine mouthwash; Drug: Oxygen
- No mouthwash and liberal oxygen during surgery (Active Comparator): No pre-surgical mouthwash in combination with 80-100% FiO2 during surgery.
  Interventions: Drug: Oxygen
- Mouthwash and restrictive oxygen during surgery (Experimental): Pre-surgical mouthwash with 0.2% chlorhexidine gluconate in combination with 21-30% FiO2 during surgery.
  Interventions: Drug: Chlorhexidine mouthwash; Drug: Oxygen
- No mouthwash and restrictive oxygen during surgery (Active Comparator): No pre-surgical mouthwash in combination with 21-30% FiO2 during surgery.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Chlorhexidine mouthwash — 0.2% Chlorhexidine digluconate
  Arms: Mouthwash and liberal oxygen during surgery; Mouthwash and restrictive oxygen during surgery
Drug: Oxygen — Oxygen 80-100%
  Arms: Mouthwash and liberal oxygen during surgery; No mouthwash and liberal oxygen during surgery
Drug: Oxygen — Oxygen 21-30 %
  Arms: Mouthwash and restrictive oxygen during surgery; No mouthwash and restrictive oxygen during surgery

SUMMARY:
PENGUIN is a pragmatic multi-center trial investigating the effects of pre-operative mouthwash and perioperative oxygen on the incidences of pneumonia and surgical site infection (SSI) following major abdominal surgery.

Patients will be recruited from low and middle income countries and randomly assigned to a trial treatment arms: a) pre-operative chlorhexidine mouthwash and 80-100% FiO2; b) no pre-operative mouthwash and 80-100% fraction of inspired oxygen (FiO2); c) pre-operative chlorhexidine mouthwash and 21- 30% FiO2; or d) no pre-operative mouthwash and 21-30% FiO2.

DETAILED DESCRIPTION:
PENGUIN is a pragmatic, blinded (outcome assessor), 2x2 factorial, multi-centre randomised controlled trial, with an internal pilot, to evaluate measures to reduce surgical site infection (SSI) and pneumonia rates in patients undergoing surgery with an abdominal incision.

Pneumonia is one of the most serious complications to occur after surgery, accounting for up to one in four of all postoperative deaths. The incidence is greater still in high-risk populations such as those undergoing midline laparotomy where mortality rates are more than 10%. SSIs are clearly important being the most frequent healthcare-associated infection in LMICs, affecting one in three patients undergoing contaminated or dirty surgery (34, 35). SSIs cause pain, discomfort and disability. They increase the time taken to return to work, and healthcare costs

The risk of postoperative mortality and complications such as surgical site infection is three times greater in low and middle-income countries (LMICs) than in high-income countries. In order to address surgical need worldwide, it is estimated that provision of a further 312 million operations would be required each year.

Patients will be recruited from hospitals in Low and Middle Income Countries (LMICs) who are undergoing elective or emergency mid-line laparotomy. Eligible patients will be randomised at the level of the individual in a 1:1:1:1 ratio between:

A. Preoperative chlorhexidine mouthwash and 80-100% FiO2 during surgery B. No preoperative chlorhexidine mouthwash and 80-100% FiO2 during surgery C. Preoperative chlorhexidine mouthwash and 21-30% FiO2 during surgery D. No preoperative chlorhexidine mouthwash and 21-30% FiO2 during surgery

The 6 month internal pilot will assess the feasibility of recruitment, compliance with treatment allocation and patient retention and follow-up rates. The main Randomised Control Trial will recruit 12,924 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children aged 10 years or over
* Elective or emergency abdominal surgery via midline laparotomy with an anticipated abdominal incision of at least 5cm in length
* Written informed consent of patient (signature or a fingerprint)

Exclusion Criteria:

* Patients undergoing caesarean section
* Patients with a documented or suspected allergy to chlorhexidine
* Patient unable to complete postoperative follow-up (not contactable after discharge)
* Previous enrolment in PENGUIN within the past 30 days
* American Society of Anesthesiologists (ASA) grade V patients (expected to die with or without surgery)

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12942 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pneumonia using the US Centers for Disease Control (CDC) definition of pneumonia (Mouthwash intervention only) | Within 30 days post-surgery from index operation
  Pneumonia will be classified using the US Centers for Disease Control (CDC) definition of pneumonia
Number of participants with surgical site infection (Oxygen therapy intervention only) | Within 30 days post-surgery from index operation
  The infection must involve the skin, subcutaneous, muscular or fascial layers of the incision AND The patient must have at least one of the following:
  * Purulent drainage from the wound
  * Organisms are detected from a wound swab
  * Wound opened spontaneously or by a clinician AND, fever (>38°C), OR at the surgical wound, the patient has at least one of: pain or tenderness; localised swelling; redness; heat;
  * Diagnosis of SSI by a clinician or radiological imaging

SECONDARY OUTCOMES:
Number of trial participant moralities (Mouthwash and oxygen therapy intervention comparisons) | Within 30 days post-surgery from index operation
  Patient mortality status
Number of participants who received repeat abdominal surgery to treat complications (Oxygen therapy intervention only) | Within 30 days post-surgery from index operation
  Repeat abdominal surgery to treat complications
Number of participants who received repeat abdominal surgery (Mouthwash and oxygen therapy interventions) | Within 30 days post-surgery from index operation
  Repeat abdominal surgery
Length of hospital stay for index admission (Mouthwash and oxygen therapy interventions) | Within 30-days post surgery from index operation
  Length of hospital stay for index admission will be collected and will measure time from surgery to time of discharge.
Number of participants returning to normal activities (Mouthwash and oxygen therapy interventions) | Within 30 days post-surgery from index operation
  Return to normal activities (e.g. work, school, or family duties) ascertained by trial specific case report forms.
Number of participants admissions to a critical care unit (Mouthwash and oxygen therapy interventions) | Within 30 days post-surgery from index operation
  Admission to a critical care unit will be captured on the trial case report forms.
Health resource usage per patient | Within 30 days post-surgery from index operation
  Resource use data will be collected as part of the economic evaluation of the different treatment combinations in a sub-group of adult patients at selected centers.
  Information related to post-operative cost (medicinal products, amenities and personal) will be collected on a health resource usage case report form designed by the trials health economist.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Pearse, Principal Investigator — Royal London Hospital
Locations (37):
- Brazil (5):
  - Hospital das Clinicas da Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Hospital Universitario Professor Edgar Santos/Bahia, Salvador
  - Hospital Sao Jose - Criciuma/SC, São José
- India (16):
  - Homi Bhabha Cancer Hospital & Research Centre, Visakhapatnam, Andhra Pradesh
  - Sher - i - Kashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir
  - Chinchpada Christian Hospital, Chinchpāda, Maharashtra
  - Kasturba Medical College Hospital, Manipal, Madhava Nagar, Manipal, Karnataka
  - Government Medical College, Patiala, Patiāla, Punjab
  - All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar
  - Government Medial College & Hospital, Chandigarh, Chandigarh
  - All India Institute of Medical Sciences, Jodhpur, Jodhpur
  - Tata Medical Center, Kolkata
  - Christian Medical College (CMC) & Hospital, Ludhiana, Ludhiana
  - Madhepura Christian Hospital, Madhepura
  - Topiwala National Medical College and Bai Yamunabai Laxman Nair Charitable Hospital, Mumbai
  - Tata Memorial Hospital, Mumbai
  - Maulana Azad Medical College, New Delhi
  - All India Institute of Medical Sciences, Rishikesh, Rishikesh
  - Christian Medical College & Hospital Vellore, Vellore
- Mexico (2):
  - Centro Médico Nacional de Occidente IMSS, Belisario Domínguez
  - Hospital Espanola Veracruz, Veracruz
- Nigeria (10):
  - University of Benin Teaching Hospital, Benin City
  - University Of Abuja Teaching Hospital, Gwagwalada
  - University College Hospital, Ibadan
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife
  - University of Ilorin Teaching Hospital, Ilorin
  - Ahmadu Bello University Teaching Hospital, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Lagos State University Teaching Hospital, Lagos
  - Lagos University Teaching Hospital, Lagos
  - Nnamdi Azikiwe University Teaching Hospital, Nnewi
- South Africa (4):
  - Tygerberg Hospital, Cape Town
  - Groote Schuur Hospital, Cape Town
  - New Somerset Hospital, Cape Town
  - Paarl Provincial Hospital, Paarl

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via a process of controlled access
Supporting Information: Study Protocol, ICF
Time Frame: 6 months post publication
Access Criteria: Formal requests must be submitted to the Data Access Group at Birmingham Clinical Trials Unit

REFERENCES:
- [Derived] PENGUIN Trial Management Groupj.glasbey@bham.ac.uk23cgeorge@gmail.com; NIHR Global Health Research Unit on Global Surgery Collaborators; PENGUIN Trial Management Group. PErioperative respiratory care aNd outcomes for patients underGoing hIgh risk abdomiNal surgery (PENGUIN): a randomised international internal pilot trial. BJA Open. 2025 Apr 10;14:100396. doi: 10.1016/j.bjao.2025.100396. eCollection 2025 Jun. PMID 40255646